CLINICAL TRIAL: NCT03942367
Title: Evaluation of the Safety and Effectiveness of the vPatch Device for the Management and Treatment of Premature Ejaculation
Brief Title: Evaluation of the Safety and Effectiveness of the vPatch Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virility Medical Ltd. (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-PR-03-01
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-07

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation; Sexual Medicine; Urology; Sexual Dysfunction
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: This is a double-blind, multi-center clinical trial. Patients enrolled will be randomized in a 2:1 ratio to receive active vPatch device (Group A) or a Sham Device (Group B).
Who Masked: Participant, Investigator
Masking Description: An unblinded sub-Investigator will preconfigure the patches to be active or sham, and pack them in 4 patches per box. The randomization will be carried out in accordance to the the instructions provided, keeping the Investigator's and Patient's blindness about the configuration of each patch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Device Group) (Experimental): Patients will receive a fully functioning vPatch device, pre-configured to deliver stimulation intensity according to the subjective motor threshold intensity reported by the Patients. Pre-configured stimulation intensity cannot be changed by the Patient.
  Interventions: Device: Active Device (vPatch)
- Group B (Sham Device Group) (Sham Comparator): Patients will receive a vPatch device pre-configured to deliver the sensory electrical stimulation according to the subjective sensory threshold that is ineffective for muscle activation. Pre-configured stimulation intensity cannot be changed by the Patient.
  Interventions: Device: Sham Device (vPatch)

INTERVENTIONS:
Device: Active Device (vPatch) — Electrical stimulation inducing motor response at the pelvic-floor muscles. Stimulation will be delivered by vPatch device configured to motor intensity.
  Arms: Group A (Active Device Group)
Device: Sham Device (vPatch) — Electrical stimulation inducing sensory response at the perineum.Stimulation will be delivered by vPatch device configured to sensory intensity.
  Arms: Group B (Sham Device Group)

SUMMARY:
Multi-center, international, prospective, randomized, double-blind, two-arms, sham-controlled, first-in-human clinical investigation.

The Patients will be allocated to one of the following groups:

* Group A (Active Device Group): Patients will receive a fully functioning vPatch device, pre-configured to deliver stimulation intensity according to the subjective motor threshold intensity reported by the Patients. Pre-configured stimulation intensity cannot be changed by the Patient.
* Group B (Sham Device Group): Patients will receive a vPatch device pre-configured to deliver the sensory electrical stimulation according to the subjective sensory threshold that is ineffective for muscle activation. Pre-configured stimulation intensity cannot be changed by the Patient.

The study will start with a Screening Visit (Visit 1), when potential Patients complaining of PE will be informed about the investigation and its objectives. If they agree to participate, after signing a valid Informed Consent Form they will undergo a full medical history and physical examination and will be selected according to eligibility criteria except IELT (which will be examined at the next visit).

The primary objective of this study is to assess the safety profile of the vPatch device and its effectiveness in delaying ejaculation when used in Patients suffering of PE.

The secondary objectives of this study are:

* To assess the Patient's perception of the ease of use of the vPatch device and treatment, through the use of a dedicated questionnaire (Usability Questionnaire).
* To assess the Patient's perception of the changes in his Premature Ejaculation Profile (PEP) under different aspects with the use of device, through the use of a dedicated questionnaire (Control and Distress Domains of the Premature Ejaculation Profile (PEP) Questionnaire).
* To assess the Patient's perceived intensity of orgasm by using the vPatch device, through the use of a validated tool (Orgasmometer).

DETAILED DESCRIPTION:
After the first visit the Patients will undergo a run-in Home Phase, during which they will be asked to have 4 sexual intercourse sessions with their female partners, in the privacy of their home, during which their partner will measure their intravaginal ejaculatory latency time (IELT) using a stopwatch.

After the run-in Home Phase the Patients will be requested to attend to the hospital (Visit 2) and the ones with a IELT value confirming their eligibility will be randomized in the trial (otherwise they will be excluded as Screening Failures).

Visit 2 will include three steps. Step 1: conditioning stimulation, delivered to the Patient's forearm muscles, aiming at familiarizing and adapting the Patient to transcutaneous electrical stimulation. Stimulation during Step 1 will be delivered using a CE approved TensMed S82 device. Following the conditioning stimulation, the Patient will undergo Step 2: incrementally increasing perineal stimulation, in order to identify the electrical intensity of his sensory and motor activation. The Patient will recognize motor activation as a muscle contraction, similarly to the voluntary induced muscle contraction when delaying urination. Step 2 will be repeated twice. Finally, the Patient will undergo Step 3: 10 to 15 minutes (according to Investigator's discretion) of continuous functional intensity stimulation, delivered to the Patient's perineum, aiming at demonstrating safety of prolonged stimulation. Stimulation during Steps 2 and 3 will be delivered using the investigational BLE (Bluetooth Low Energy)-enabled vPatch device. Furthermore, the Investigator will carefully instruct the Patient how to safely place the device, how to safely use of the device, and how to remove the device. During this visit the baseline assessments (see flow chart) will be carried out.

Following the Visit 2, the Home Phase will initiate, where the Patients will be asked to have 4 sexual intercourse sessions with their female partners, in the privacy of their home, during which their partner will measure their Intravaginal Ejaculatory Latency Time (IELT) using a stopwatch. The 4 sessions will include four IELT measurements, while the investigational BLE-disabled vPatch device is applied, pre-configured either delivering a functional stimulation to 40 Patients (Active Device Group) or sensory stimulation to 20 Patients (Sham Device Group). All Patients will be informed that the stimulation is not necessarily detectable. The Investigator will call the Patients every day during the first three days of the Home Phase to monitor the progression and to remind to fill in the 72 h Safety Questionnaire.

The Patients will be requested to return to the site (Visit 3) after 4 intercourse sessions with their female partners in order to undergo the assessments foreseen by protocol (see flow chart) and to return the filled questionnaires and the used device. This will be considered the End of Trial Visit.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male Patients, aged ≥ 18 and ≤ 60 years old.
2. Patients who are diagnosed with clinical premature ejaculation or with self-perceived ELT < 3 minutes.
3. Patients with stable, heterosexual, monogamous, sexual relationship for at least 3 months at the time of the enrolment.
4. Patients planning to maintain the relationship for the whole duration of the study.
5. Patients with 75% of IELT baseline measurement < 2 minutes and 25% of IELT baseline measurement < 3 minutes at Visit 2.
6. Patients with PEDT (Premature Ejaculation Diagnostic Tool) measurement ≥ 11 at the time of enrolment.
7. Patients with IIEF-5 (International Index of Erectile Function) measurement ≥ 22 at the time of enrolment.
8. Patients understanding the nature of the study and providing their informed consent to participation.
9. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol.

EXCLUSION CRITERIA:

1. Patients with history of cardiovascular disorders.
2. Patients with history of other sexual dysfunction (other than PE).
3. Patients suffering of erectile dysfunction.
4. Patients carrying any type of implanted pacemaker/defibrillator.
5. Patients suffering of diagnosed Diabetes Mellitus with peripheral neuropathy.
6. Patients suffering of perineal dermatological diseases.
7. Patients suffering of perineal skin irritation / lesions.
8. Patients suffering of any psychiatric major disease (axis 1) and/or taking any relevant medications.
9. Patients taking antidepressant therapy, topical anesthetic agents or sexual-related cognitive behavioral therapy within the 4 weeks before the enrolment.
10. Patients with past occurrences of ejaculation before intromission.
11. Patients with history of genital or anorectal neoplastic illness in the 2 years before the enrolment.
12. Patients with pregnant partner.
13. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
14. Patients with any medical incidence where the use of the device may jeopardize the Patient's safety per Investigator's discretion.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male Patients, aged ≥ 18 and ≤ 60 years old.
Enrollment: 59 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Adverse events rate during the study period. All adverse occurrences (serious/non-serious or device-related/non device-related) will be recorded prospectively, categorized and evaluated for causality using defined criteria. | Entire Study Period (up to 2,5 months)
  Primary Endpoint of Safety
Objective: change in IELT from baseline (V2) to the end of Home Phase Visit (V3). | Up to 56 days
  Primary Endpoint of Device Performance
Subjective: proportion of patients reporting an improvement according to the Clinical Global Impression of Change (CGIC) measured at V3. | Up to 56 days
  Primary Endpoint of Device Performance

SECONDARY OUTCOMES:
Evaluation of Patient's subjective outcome assessment of the Premature Ejaculation Profile (PEP) from baseline (V2) to the end of Home Phase Visit (V3). | Up to 56 days
  Secondary Endpoint of Device Performance
Evaluation of Patient's subjective outcome assessment of orgasmic intensity via Orgasmometer from baseline (V2) to the end of Home Phase Visit (V3). | Up to 56 days
  Secondary Endpoint of Device Performance
Evaluation of Patient's subjective outcome assessment of ease of use of the vPatch device and treatment during Home Phase. | Entire Study Period (up to 2,5 months)
  Secondary Endpoint of Device Performance

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Sexual Dysfunction Clinic, Rambam Medical Center - Haifa, Israel
Locations (3):
- Sexual Dysfunction Clinic, Rambam Medical Center, Haifa, Israel
- Italy (2):
  - Urologia, Casa di Cura "Villa Donatello", Sesto Fiorentino, Firenze
  - U.O.C. Urologia e Centro di litotrissia urinaria D.A.I. Nefrologia, urologia e chirurgia generale e dei trapianti di rene, anestesia e rianimazione, A.O.U. "Federico II" di Napoli, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giuliano F, Patrick DL, Porst H, La Pera G, Kokoszka A, Merchant S, Rothman M, Gagnon DD, Polverejan E; 3004 Study Group. Premature ejaculation: results from a five-country European observational study. Eur Urol. 2008 May;53(5):1048-57. doi: 10.1016/j.eururo.2007.10.015. Epub 2007 Oct 16. PMID 17950985
- [Background] Tang WS, Khoo EM. Prevalence and correlates of premature ejaculation in a primary care setting: a preliminary cross-sectional study. J Sex Med. 2011 Jul;8(7):2071-8. doi: 10.1111/j.1743-6109.2011.02280.x. Epub 2011 Apr 14. PMID 21492404
- [Background] Althof SE. Prevalence, characteristics and implications of premature ejaculation/rapid ejaculation. J Urol. 2006 Mar;175(3 Pt 1):842-8. doi: 10.1016/S0022-5347(05)00341-1. PMID 16469562
- [Background] Shafik A. The mechanism of ejaculation: the glans-vasal and urethromuscular reflexes. Arch Androl. 1998 Sep-Oct;41(2):71-8. doi: 10.3109/01485019808987948. PMID 9730435
- [Background] Dinsmore WW, Hackett G, Goldmeier D, Waldinger M, Dean J, Wright P, Callander M, Wylie K, Novak C, Keywood C, Heath P, Wyllie M. Topical eutectic mixture for premature ejaculation (TEMPE): a novel aerosol-delivery form of lidocaine-prilocaine for treating premature ejaculation. BJU Int. 2007 Feb;99(2):369-75. doi: 10.1111/j.1464-410X.2006.06583.x. Epub 2006 Nov 24. PMID 17129234
- [Background] Patrick DL, Giuliano F, Ho KF, Gagnon DD, McNulty P, Rothman M. The Premature Ejaculation Profile: validation of self-reported outcome measures for research and practice. BJU Int. 2009 Feb;103(3):358-64. doi: 10.1111/j.1464-410X.2008.08041.x. Epub 2008 Sep 12. PMID 18793300
- [Background] Althof SE, Brock GB, Rosen RC, Rowland DL, Aquilina JW, Rothman M, Tesfaye F, Bull S. Validity of the patient-reported Clinical Global Impression of Change as a measure of treatment response in men with premature ejaculation. J Sex Med. 2010 Jun;7(6):2243-2252. doi: 10.1111/j.1743-6109.2010.01793.x. Epub 2010 Mar 30. PMID 20367770
- [Background] Limoncin E, Lotti F, Rossi M, Maseroli E, Gravina GL, Ciocca G, Mollaioli D, Di Sante S, Maggi M, Lenzi A, Jannini EA. The impact of premature ejaculation on the subjective perception of orgasmic intensity: validation and standardisation of the 'Orgasmometer'. Andrology. 2016 Sep;4(5):921-6. doi: 10.1111/andr.12220. Epub 2016 May 23. PMID 27214119
- [Derived] Shechter A, Mondaini N, Serefoglu EC, Gollan T, Deutsch F, Appel B, Gruenwald I. A novel on-demand therapy for lifelong premature ejaculation using a miniature transperineal electrical stimulator-the vPatch: an as-treated analysis. J Sex Med. 2023 Jan 14;20(1):22-29. doi: 10.1093/jsxmed/qdac012. PMID 36897239
- See also: Virility Medical Ltd. official website — https://www.virilitymedical.com/